CLINICAL TRIAL: NCT01439555
Title: Endothelial Facilitation in Alzheimer's Disease. An Open Label Pilot Study of the Sequential and Cumulative Effects of Simvastatin, L-Arginine, and Sapropterin (Kuvan) on Cerebral Blood Flow and Cognitive Function in Patients With Alzheimer's Disease.
Brief Title: Endothelial Facilitation in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: The Glass Foundation (Unknown)
Responsible Party: Principal Investigator, Elizabeth Degrush, Assistant Professor, Psychiatry, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13748
Record Dates: First submitted 2011-09-16; First posted 2011-09-23 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Alzheimer's Disease
Keywords: Early Alzheimer; Mild Cognitive Impairment; Drug treatment; Cerebral blood flow; Endothelial facilitation; Cognitive improvement
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Simvastatin; sapropterin; Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Simvastatin + L-Arginine + Tetrahydrobiopterin (Experimental): Simvastatin, 40 mg per day orally; L-Arginine, 2 Gm four times per day orally; Tetrahydrobiopterin 20 mg/kg/day orally
  Interventions: Drug: Simvastatin; Drug: L-Arginine; Drug: Tetrahydrobiopterin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin, 40 mg per day orally
  Other Names: Tetrahydrobiopterin
Drug: L-Arginine — L-Arginine, 2 Gm four times per day orally;
Drug: Tetrahydrobiopterin — Tetrahydrobiopterin 20 mg/kg/day orally
  Other Names: Kuvan; Sapropterin

SUMMARY:
Purpose of the study: Patients with mild Alzheimer's Disease will be given three different drugs over a 4-month period to try to increase the blood flow to their brains, and improve blood vessel and brain function. Each drug can help to open the blood vessels in the brain, and together they may be more effective than each drug alone. The hypothesis is that small blood vessels secrete substances that maintain the integrity of the brain, and may prevent loss of nerve cells leading to Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have mild Alzheimer's Disease or Mild Cognitive Impairment (MCI);
* age between 55-85;
* Mini Mental Status Exam (MMSE) between 15-26;
* a caregiver who can provide information, and bring patient to the sessions;
* no known allergies to any of the medications to be used;
* normal renal function; willingness of patient and spouse/responsible caregiver to participate.

Exclusion Criteria:

* Significant Psychiatric disorder;
* stroke; current use of any of the test medications (e.g., statin, L-Arginine, Kuvan);
* phenylketonuria (PKU) ;
* elevated serum phenylalanine level (>10 mg/dL);
* allergy to any of the medications; current active malignancy;
* renal insufficiency (elevated creatinine above 1.3mg/dl);
* abnormal liver function (Alanine Aminotransferase (ALT) or Aspartate Transaminase (AST) 2x normal);
* other serious disease including coronary insufficiency or congestive heart failure, carotid stenosis greater than 50%, active peptic ulcer, urinary tract or other active infection, cancer (except skin cancer, or 5 years inactive breast or prostate cancer )etc.;
* pregnancy; or
* inability to come to UMass for follow-up. Subjects may continue to take anticholinesterase drugs for Alzheimer's Disease (Aricept, Exelon, Razadyne) and/or Namenda, if they have been on the drug(s) for at least 3 months. Subjects on levodopa and male subjects taking drugs for erectile dysfunction (Viagra, Cialis, Levitra) are cautioned regarding hypotension.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R DeGrush, DO, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School/ UMass Memorial Medical Center, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Degrush E, Shazeeb MS, Drachman D, Vardar Z, Lindsay C, Gounis MJ, Henninger N. Cumulative effect of simvastatin, L-arginine, and tetrahydrobiopterin on cerebral blood flow and cognitive function in Alzheimer's disease. Alzheimers Res Ther. 2022 Sep 17;14(1):134. doi: 10.1186/s13195-022-01076-7. PMID 36115980

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
Started | 11
Completed | 10
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Prospective, open-label, single group assignment, single center study conducted by UMass Medical School at the UMass Memorial Medical Center in Worcester, MA. 11 subjects total were screened and enrolled in this study, 10 subjects completed the study as 1 subject was initially enrolled but was excluded due to not meeting inclusion criteria.
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: Years of Age] | 67.1 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Cerebral Blood Flow as Measured by Magnetic Resonance Imaging (MRI)
Description: Measurement of changes to cerebral blood flow (ml/110g/min) in regions of interest as measured using Magnetic Resonance Imaging (MRI)
Time Frame: Baseline to 16 weeks
Population: Data for 6 participants available. Data file for remaining participants corrupted and could not be retrieved for analysis/reporting.
Measure: Mean (Standard Deviation); unit: ml/110g/min
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
Number analyzed (Participants) | 6
ml/110g/min
  Baseline | 0.621528 (0.116513988)
  Week 4 | 0.6447692 (0.070388324)
  Week 8 | 0.654822667 (0.024032403)
  Week 16 | 0.579838667 (0.091658076)

2. Primary Outcome: Change in Cerebral Blood Flow as Measured by Arterial Spin Labeling During Magnetic Resonance Imaging (MRI)
Description: Data not available as files corrupted and could not be analyzed
Time Frame: Baseline to week 16
Population: Data files corrupted, analysis not possible
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
Number analyzed (Participants) | 0

3. Secondary Outcome: Mini Mental State Examination (MMSE) Scores
Description: Change in mental state as reflected by changes to mean Mini Mental State Examination (MMSE) score as measured 4 weeks, 8 weeks and 16 weeks post-baseline. The MMSE uses a 30 point questionnaire to measure cognitive impairment. The MMSE is scored from 0 to 30,with a score equal to or greater than 24 points indicating normal cognition, a score of 19-23 points indicating mild cognitive impairment, 10-18 points indicating moderate impairment and a score equal to or below 9 indicating severe impairment.
Time Frame: Baseline to 4 weeks, 8 weeks and 16 weeks post-baseline
Population: Patients were sequentially treated with the HMC-CoA reductase synthesis inhibitor simvastatin (weeks 0-16); L-Arginine (weeks 4-16); and tetrahydrobiopterin (weeks 8-16). The investigators assessed cognitive function with a psychometric battery including the MMSE at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
Number analyzed (Participants) | 10
score on a scale
  Baseline | 24.2 (3.155)
  Week 4 | 25.33 (2.21)
  Week 8 | 26 (3.13)
  Week 16 | 25.55 (2.51)

4. Secondary Outcome: Cognitive Assessment Screening Test (CAST)
Description: This outcome measured the change in average Cognitive Assessment Screening Test (CAST) scores for the participant group. The CAST is scored from 0 to 40. A higher score indicates better performance, and a lower score indicates worse performance. The participants were given the CAST at baseline, 4 weeks, 8 weeks and 16 weeks post-baseline. The outcome reports on the averaged change for the averaged CAST scores from baseline to 16 weeks.
Time Frame: Baseline to 16 weeks post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
Number analyzed (Participants) | 10
score on a scale | 31.4 (5.46)

5. Secondary Outcome: Clinical Dementia Rating Scale (CDR)
Description: This outcome measures Clinical Dementia Rating Scale (CDR) scores at baseline (enrollment) and 16 weeks post-enrollment. The Clinical Dementia Rating Scale is scored with a composite scale of 0 to 3, with higher scores indicating lower functional status and lower scores indicating better functional status.
Time Frame: Baseline to 16 weeks post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
Number analyzed (Participants) | 10
score on a scale
  CDR Score at Baseline | 0.9 (.47)
  CDR Score at 16 weeks | 0.9 (.47)

6. Secondary Outcome: Alzheimer's Disease Assessment Scale: Cognitive and Modified Version (ADAS-COG)
Description: Mean Alzheimer's Disease Assessment Scale: Cognitive Subscale (ADAS-COG) score at baseline and at 16 weeks post-enrollment. The ADAS-COG consists of 11 tasks measuring disturbances of memory, language, praxis, attention and other cognitive abilities. Total scores range from 0 to 70, with higher scores (18 and above) indicating greater cognitive impairment.
Time Frame: Baseline to 16 weeks post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
Number analyzed (Participants) | 10
score on a scale
  ADAS-COG Baseline | 21.6 (5.65)
  ADAS-COG 16 weeks | 21.9 (8.9)

7. Secondary Outcome: Clinical Interview Based Impression of Change + Caregiver Input (CIBIC Plus)
Description: The Clinical Interview Based Impression of Change + Caregiver Input (CIBIC Plus) is a semi-structured instrument to examine four major areas of patient function: General, Cognitive, Behavioral and Activities of Daily Living. It is scored from 1 to 7. A score of 1 indicates marked improvement, 4 indicates no change and 7 indicates marked worsening.
Time Frame: Baseline to 4 weeks, 8 weeks and 16 weeks post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
Number analyzed (Participants) | 10
score on a scale
  Change in CIBIC score from baseline to 4 weeks | -.1 (0.32)
  Change in CIBIC Score from 4 weeks to 8 weeks | .6 (.84)
  Change in CIBIC Score from 8 weeks to 16 weeks | -.1 (1.29)

ADVERSE EVENTS:
Time Frame: 6 Years.
Arm/Group | Simvastatin + L-Arginine + Tetrahydrobiopterin
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
The data for the MRI measurements (cerebral blood flow) experienced file corruption, rendering segments of data irretrievable and the whole set non-analyzable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT01439555/Prot_SAP_000.pdf